CLINICAL TRIAL: NCT06737952
Title: Cellular and Molecular Analysis of Synovial Tissue of Patients With Arthritis
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: 2024-02011; mu24kyburz
Record Dates: First submitted 2024-12-11; First posted 2024-12-17 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Arthritis; Arthritis, Rheumatoid; Osteoarthritis; Spondyloarthritis; Synovitis
Keywords: ultrasound-guided synovial biopsies (UGSB); inflammatory response; synovial biopsy
MeSH Terms: conditions — Arthritis; Arthritis, Rheumatoid; Osteoarthritis; Spondylarthritis; Synovitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Days
Biospecimen Retention: Samples With DNA — * Synovial tissue samples collected from inflamed joints, samples at least 6 mm in size with typical characteristics of synovium
  * Synovial fluid
  * peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to study the inflammatory response in various forms of arthritis.

DETAILED DESCRIPTION:
Arthritis, a significant heald burden is characterized by joint inflammation that severely impacts patients' quality of live. Despite advancements in treatment, many individuals with conditions like rheumatoid arthritis (RA), osteoarthritis (OA), and spondyloarthritis (SpA) do not achieve satisfactory outcomes, underscoring the need for more precise therapeutic strategies.

The project aims to characterize the inflammatory response in various form of arthritis by collecting and analyzing synovial tissue-the connective tissue lining joints. Biopsies will be collected through ultrasound-guided biopsies (UGSB), a minimally invasive and well-tolerated procedure. Presence of immune and stromal cells in the tissue, their interactions, and their relationship to clinical symptoms are characterized by histological and molecular methods. By comparing these features across different forms of arthritis, the study aims to identify molecular pathways and biomarkers that distinguish these diseases and their subtypes. The study hopes to contribute to a broader understanding of arthritis pathophysiology, ultimately translating into novel therapeutic targets and tailored clinical strategies.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Clinically relevant arthritis in one or more joints as assessed by the treating rheumatologist, including RA, SpA, connective tissue disease and OA.

Exclusion Criteria:

* Known allergies to local anesthetics
* Family history of bleeding, history of increased bleeding tendency or prolonged bleeding, current treatment with oral anticoagulants or platelet aggregation inhibitors; Quick < 65%, international normalised ratio (INR) ≥ 1.3, thrombocyte count < 100'000/μl, activated partial thromboplastin time (aPTT) > 37 sec
* Inability or insufficient knowledge of project language to understand the information given in the informed consent form

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: arthritis patients
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2029-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Grade of synovitis | immediately after collection to study completion, up to 5 years
  assessed by the Krenn score in the hematoxylin and eosin staining (Score 0-3, 0=normal, 3=severe)
classification pathotypes | immediately after collection to study completion, up to 5 years
  immunohistochemical staining with cell type specific markers including CD15, CD68, CD3, CD20, CD138 of the collected tissues from different arthritis subtypes
comparing transcriptomic signature | immediately after collection to study completion, up to 5 years
  single-cell RNA sequencing of collected tissues from different arthritis subtypes to identify disease specific biomarkers.

CONTACTS AND LOCATIONS:
Overall Officials: Diego Kyburz, Prof. Dr., Principal Investigator — Universitätsspital Basel